CLINICAL TRIAL: NCT04897477
Title: An Open Label, Single Arm, Phase I/II in the Combination of Azacytidine, Bendamustine and Piamprizumab in Refractory/Relapsed B-cell Non-Hodgkin's
Brief Title: Azacytidine, Bendamustine, Piamprizumab in Refractory/Relapsed B-cell Non-Hodgkin's Lymphoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Han weidong, Professor, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PLAGH-BT-066
Record Dates: First submitted 2021-05-18; First posted 2021-05-21 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Non-hodgkin Lymphoma,B Cell
MeSH Terms: interventions — Azacitidine; Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- combination of Azacytidine, Bendamustine and Piamprizumab (Experimental): combination of Azacytidine, Bendamustine and Piamprizumab in Refractory/Relapsed B-cell Non-Hodgkin's Lymphoma, every 28 days
  Interventions: Drug: Azacytidine, Bendamustine and Piamprizumab

INTERVENTIONS:
Drug: Azacytidine, Bendamustine and Piamprizumab — Azacytidine by means of subcutaneous injection, Bendamustine and Piamprizumab intravenous infusion

SUMMARY:
This is an open label, single arm, phase I/II for patients with r/r Non-Hodgkin's Lymphoma

. The purpose is to evaluate the safety and efficacy of the combination with Azacytidine, Bendamustine and Piamprizumab

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 and ≤80 years
2. Performance status (ECOG) between 0 and 3.
3. Histologically confirmed B-cell non-Hodgkin lymphoma (NHL), including the following types defined by WHO 2016.
4. Refractory disease or relapsed after treatment with ≥2 lines of chemotherapy and either having failed autologous HSCT or being ineligible for or not consenting to autologous HSCT; or not suitable for CAR T treatment or resistance, progression or relapse after CAR T treatment; or CAR T pre-culturing losers can also be enrolled.
5. Adequate organ function.
6. An adequate bone marrow reserve.
7. Measurable or assessable disease according to the"IWG Response Criteria for Malignant Lymphoma"(Cheson 2014). Patients in complete remission (CR) with no evidence of disease were not eligible.
8. Informed consent/assent requiring that all patients have the ability to understand and the willingness to provide written informed consent.
9. Life expectancy > 12 weeks.
10. Patients with definite involvement of the gastrointestinal tract, and patients with central nervous system (CNS) by PETCT and MRI involvement were allowed to enrolled in this clinical study.

Exclusion Criteria:

1. Pregnant or lactating women.
2. Uncontrolled medical disorders, active bacterial, viral infection or treponema pallidum infection and so on.
3. Requirement for urgent therapy due to tumor mass effects such as respiratory obstruction or blood vessel compression.
4. Current or expected need for systemic corticosteroid therapy.
5. Any organ failure.
6. Patients with a second tumor requiring therapy or intervention.
7. Subjects considered unlikely to complete all protocol-required study visits or procedures, including follow-up visits, or comply with the study requirements for participation according to the investigator's judgement.
8. Prior organ allograft.
9. Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-04-22 (Actual); Primary Completion 2022-04-23 (Estimated); Study Completion 2023-04-23 (Estimated)

PRIMARY OUTCOMES:
Safety: treatment-related adverse events (AEs) | 6 month
  Incidence, nature, and severity of adverse events graded according to the NCI CTCAE v5.0. AEs were considered to be treatment-related if they had started or worsened within the interval from first study drug administration until the follow-up visit.

SECONDARY OUTCOMES:
Objective Response Rate | 6 month
  The ORR is defined as the proportion of patients with a best overall disease response, including complete response (CR) and partial response (PR).
Complete Response Rate | 6 month
  CR rate assess by investigators per the 2014 Lugano classification rate of subjects achieved complete response in all evaluable subjects

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Biotherapeutic Department of Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Biotherapeutic Department of Chinese PLA General Hospital, Beijing